CLINICAL TRIAL: NCT03014856
Title: Identification of Metabolic Phenotypes in Childhood Obesity by 1H-NMR Metabolomics of Blood Plasma
Brief Title: Metabolic Phenotypes in Childhood Obesity
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Peter Adriaensens, Professor (hoogleraar), Hasselt University
Other Study IDs: LCRP-OBNMR
Record Dates: First submitted 2016-12-13; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Obesity, Pediatric
Keywords: Metabolic syndrome; Metabolomics; NMR spectroscopy
MeSH Terms: conditions — Pediatric Obesity; Metabolic Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma for proton-NMR spectroscopy

GROUPS / COHORTS (2):
- OB-NMR: overweight and obese children and adolescents
  Interventions: Other: Blood sampling
- NMR-C: normal-weight children and adolescents
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Determine the metabolic phenotype of blood plasma by proton-NMR spectroscopy

SUMMARY:
This study provides a sound basis towards a better understanding of the biochemical mechanisms behind childhood obesity and its metabolic phenotypes, which will be of great importance towards the development of more personalized prevention and treatment in future.

DETAILED DESCRIPTION:
The aim of this study was to identify the plasma metabolic profile associated with childhood obesity and its phenotypes..

This cross-sectional study was set-up to examine the metabolic profile in fasting plasma samples from 65 overweight and obese (OB) children and 37 normal-weight (NW) controls aged 8 to 18 years. The obtained plasma 1H-NMR spectra were rationally divided into 110 integration regions, representing the metabolic phenotype. These integration regions reflect the relative metabolite concentrations and were used as statistical variables to construct a classification model in discriminating between OB and NW children and adolescents. In addition, two metabolic phenotypes were defined within the OB group, i.e. the metabolically "healthy" obese (MHO) and metabolically unhealthy obese (MUO) phenotype which are both classified as obese but with respectively, none (MHO) or at least two components (MUO) of the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* aged 8 to 18
* normal-weight, overweight or obese according to the International Obesity Task Force (IOTF) Body Mass Index (BMI) criteria
* fasted for at least 8 hours

Exclusion Criteria:

* Subjects taking any medication or having serious chronic or acute illness within two weeks preceding the clinical examination,

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 65 overweight and obese (OB) children and 37 normal-weight (NW) controls aged 8 to 18 years
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
metabolic phenotype of childhood obesity | day 1
  Significant metabolic changes in blood plasma of obese children and adolescents and normal-weight control subjects

SECONDARY OUTCOMES:
metabolic phenotype of metabolically healthy and unhealthy obese children and adolescents | day 1
  Significant metabolic changes in blood plasma of metabolically healthy obese and metabolically unhealthy obese children and adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Peter Adriaensens, PhD, Principal Investigator — Institute of Material Research, Hasselt University; Liene Bervoets, PhD, Study Chair — Hasselt University; Guy Massa, PhD, MD, Study Chair — Jessa Ziekenhuis Hasselt; Wanda Guedens, PhD, Study Chair — Institute of Material Research, Hasselt University; Gunter Reekmans, Ing, Study Chair — Institute of Material Research, Hasselt University; Jean-Paul Noben, PhD, Study Chair — BIOMED, Hasselt University

REFERENCES:
- [Background] Beckonert O, Keun HC, Ebbels TM, Bundy J, Holmes E, Lindon JC, Nicholson JK. Metabolic profiling, metabolomic and metabonomic procedures for NMR spectroscopy of urine, plasma, serum and tissue extracts. Nat Protoc. 2007;2(11):2692-703. doi: 10.1038/nprot.2007.376. PMID 18007604
- [Background] Prince RL, Kuk JL, Ambler KA, Dhaliwal J, Ball GD. Predictors of metabolically healthy obesity in children. Diabetes Care. 2014 May;37(5):1462-8. doi: 10.2337/dc13-1697. Epub 2014 Feb 26. PMID 24574347
- [Background] Butte NF, Liu Y, Zakeri IF, Mohney RP, Mehta N, Voruganti VS, Goring H, Cole SA, Comuzzie AG. Global metabolomic profiling targeting childhood obesity in the Hispanic population. Am J Clin Nutr. 2015 Aug;102(2):256-67. doi: 10.3945/ajcn.115.111872. Epub 2015 Jun 17. PMID 26085512
- [Background] Perng W, Gillman MW, Fleisch AF, Michalek RD, Watkins SM, Isganaitis E, Patti ME, Oken E. Metabolomic profiles and childhood obesity. Obesity (Silver Spring). 2014 Dec;22(12):2570-8. doi: 10.1002/oby.20901. Epub 2014 Sep 24. PMID 25251340
- [Background] Mihalik SJ, Michaliszyn SF, de las Heras J, Bacha F, Lee S, Chace DH, DeJesus VR, Vockley J, Arslanian SA. Metabolomic profiling of fatty acid and amino acid metabolism in youth with obesity and type 2 diabetes: evidence for enhanced mitochondrial oxidation. Diabetes Care. 2012 Mar;35(3):605-11. doi: 10.2337/DC11-1577. Epub 2012 Jan 20. PMID 22266733
- [Background] Wahl S, Yu Z, Kleber M, Singmann P, Holzapfel C, He Y, Mittelstrass K, Polonikov A, Prehn C, Romisch-Margl W, Adamski J, Suhre K, Grallert H, Illig T, Wang-Sattler R, Reinehr T. Childhood obesity is associated with changes in the serum metabolite profile. Obes Facts. 2012;5(5):660-70. doi: 10.1159/000343204. Epub 2012 Oct 4. PMID 23108202
- [Derived] Bervoets L, Massa G, Guedens W, Reekmans G, Noben JP, Adriaensens P. Identification of metabolic phenotypes in childhood obesity by 1H NMR metabolomics of blood plasma. Future Sci OA. 2018 May 23;4(6):FSO310. doi: 10.4155/fsoa-2017-0146. eCollection 2018 Jul. PMID 30057787